CLINICAL TRIAL: NCT01530126
Title: Platelet Derived Growth Factor Stimulates Bone Fill and Rate of Attachment Level Gain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Responsible Party: Principal Investigator, William Giannobile, Principal Investigator, University of Michigan
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2005 - PDGF
Record Dates: First submitted 2012-02-06; First posted 2012-02-09 (Estimated); Last update posted 2016-01-08 (Estimated); Status verified 2016-01

CONDITIONS: Periodontitis
Keywords: periodontitis
MeSH Terms: conditions — Periodontitis | interventions — Becaplermin; Buffers

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- B-TCP +buffer (Active Comparator): Administration of synthetic beta-tricalcium phosphate (B-TCP) mixed in sodium acetate buffer only.
  Interventions: Biological: B-TCP +buffer
- B-TCP + 0.3 mg/ml rhPDGF-BB in buffer (Experimental): Administration of synthetic beta-tricalcium phosphate (B-TCP) mixed with purified 0.3 mg/ml recombinant human platelet-derived growth factor (rhPDGF-BB) in sodium acetate buffer.
  Interventions: Biological: B-TCP + 0.3 mg/ml rhPDGF-BB in buffer
- B-TCP + 1.0 mg/ml rhPDGF-BB in buffer (Experimental): Administration of synthetic beta-tricalcium phosphate (B-TCP) mixed with purified 1.0 mg/ml recombinant human platelet-derived growth factor (rhPDGF-BB) in sodium acetate buffer.
  Interventions: Biological: B-TCP + 1.0 mg/ml rhPDGF-BB in buffer

INTERVENTIONS:
Biological: B-TCP + 0.3 mg/ml rhPDGF-BB in buffer — B-TCP mixed with sodium acetate buffer and 0.3 mg/ml rhPDGF-BB and placed into osseous defect once at baseline visit.
  Arms: B-TCP + 0.3 mg/ml rhPDGF-BB in buffer
Biological: B-TCP + 1.0 mg/ml rhPDGF-BB in buffer — B-TCP mixed with sodium acetate buffer and 1.0 mg/ml rhPDGF-BB and placed into osseous defect once at baseline visit.
  Arms: B-TCP + 1.0 mg/ml rhPDGF-BB in buffer
Biological: B-TCP +buffer — B-TCP mixed with sodium acetate buffer and placed into osseous defect once at baseline visit.
  Arms: B-TCP +buffer

SUMMARY:
The aim of the study was to evaluate the safety and effectiveness of Platelet Derived Growth Factor (PDGF) mixed with b tricalcium phosphate (BTCP) for the treatment of advanced periodontal osseous defects at 6 months of healing.

DETAILED DESCRIPTION:
This triple blind, prospective and parallel arm trial was conducted in subjects requiring surgical treatment of a periodontal osseous defect.

ELIGIBILITY:
Inclusion Criteria:

* probing depth of 7mm or greater at baseline
* following debridement, 4mm or greater vertical bone defect depth with at least one intact bony wall
* sufficient keratinized tissue to allow complete tissue coverage of the defect
* a radiographic base of the defect at least 3mm coronal to the apex of the tooth
* no evidence of localized aggressive periodontitis
* smoke less than 1 pack of cigarettes per day

Exclusion Criteria:

* failure to maintain adequate oral hygiene
* pregnant women or women intending to become pregnant
* history of oral cancer within last 6 months or HIV
* history within last year of periodontal surgery on study tooth
* study tooth mobility greater than 2
* study tooth exhibiting a class 3 furcation defect
* signs of untreated acute infection at the surgical site, apical pathology, root fracture, severe root irregularities, cemental pearls, cementoenamel junction (CEJ) projections not easily removed, untreated carious lesions at the CEJ or on the root surface, subgingival restorations or restorations with open margins at or below CEJ
* history within 6 months of weekly or more frequent use of smokeless chewing tobacco, pipe or cigar smoking, or more than 20 cigarettes a day
* allergy to yeast derived products
* investigational therapy within 30 days of surgery

Ages: 25 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Actual)
Dates: Start 2000-01; Primary Completion 2005-01 (Actual); Study Completion 2007-01 (Actual)

PRIMARY OUTCOMES:
Rate of CAL Gain | Baseline to 6 months
  Measurements for the rate of clinical attachment levels (CAL)

SECONDARY OUTCOMES:
Change in Gingival Recession (GR) | Baseline to 6 months
  Measurements in changes of gingival recession (GR)

CONTACTS AND LOCATIONS:
Overall Officials: William Giannobile, DDS, DMedSc, Principal Investigator — University of Michigan
Locations (1):
- University of Michigan School of Dentistry, Ann Arbor, Michigan, United States

REFERENCES:
- [Result] Nevins M, Giannobile WV, McGuire MK, Kao RT, Mellonig JT, Hinrichs JE, McAllister BS, Murphy KS, McClain PK, Nevins ML, Paquette DW, Han TJ, Reddy MS, Lavin PT, Genco RJ, Lynch SE. Platelet-derived growth factor stimulates bone fill and rate of attachment level gain: results of a large multicenter randomized controlled trial. J Periodontol. 2005 Dec;76(12):2205-15. doi: 10.1902/jop.2005.76.12.2205. PMID 16332231
- [Result] Nevins M, Kao RT, McGuire MK, McClain PK, Hinrichs JE, McAllister BS, Reddy MS, Nevins ML, Genco RJ, Lynch SE, Giannobile WV. Platelet-derived growth factor promotes periodontal regeneration in localized osseous defects: 36-month extension results from a randomized, controlled, double-masked clinical trial. J Periodontol. 2013 Apr;84(4):456-64. doi: 10.1902/jop.2012.120141. Epub 2012 May 21. PMID 22612364